CLINICAL TRIAL: NCT01747603
Title: The GROWNDUP Study: Pilot to Assess the Feasibility of an RCT for Promoting Growth, Nutrition and Development Through a Specialized Late Preterm Clinic
Brief Title: The GROWNDUP Study of Late Preterm Births
Acronym: GROWNDUP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-156
Record Dates: First submitted 2012-12-03; First posted 2012-12-11 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Preterm Birth
Keywords: Late preterm infant; Complications; Hospital readmissions; Follow-up; Pilot study
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Current management of LPTB (No Intervention): The current pragmatic, but non-systematic, pattern of management of LPTB infants. Growth measurements, feeding histories/methods, illness history including emergent visits to clinicians, walk-in clinics and emergency departments and breast-feeding support clinics, and basic developmental milestones (as itemized in the Rourke Developmental screening tool) will be recorded by families and primary health care providers as itemized in the Memory Book at the assessments made at the discretion of the health care providers.
- Specialized LPTB Clinic (Experimental): Additional 6 specialized LPTB follow-up clinic visits attended by pediatricians and neonatologists. Detailed findings from physical examination, feeding histories/methods, illness history including emergent visits to clinicians, walk-in clinics and emergency departments and breast-feeding support clinics, basic developmental milestones (as itemized in the Rourke Developmental screening tool) and physician recommendations will be recorded at each appointment. These will be compared to those obtained from families and primary health care providers as itemized in the Memory Book.
  Interventions: Other: Specialized LPTB clinic

INTERVENTIONS:
Other: Specialized LPTB clinic — 50% of enrolled infants will be randomized to the specialized LPTB follow-up clinic.
  Arms: Specialized LPTB Clinic

SUMMARY:
This pilot study will examine the feasibility of conducting a large randomized clinical trial (RCT) to examine the role of a novel, specialized follow-up clinic in preventing complications among late preterm infants (LPTB), born between 34 and 36 weeks gestational age. 1) Study Process: Success will be achieved if 80% of a target population of 100 subjects is met within the first 6 months of recruitment being initiated. 2) Study Resources: Success will be achieved if 80% of follow up appointments are scheduled in a timely manner and if specialized LPTB physicians in the intervention complete assessments 75% of the time in the allocated time frame and 3) Scientific: 95% data completeness on data collection forms will be identified as success

A specialized LPTB follow-up clinic is innovative as no studies have evaluated such a programme and standardized follow-up and guidelines for the care of LPTB infants after discharge from hospital do not exist. Until recently, the incorrect assumption has been that these infants are healthy and have limited risks compared to term infants.

The study's main question, in addition to assessing the feasibility of this pilot, is: "Do differences exist in short-tem clinical and developmental outcomes among LPTB infants enrolled in an RCT who are randomized to a specialized LPTB follow-up programme when compared to infants randomized to current pragmatic management?" A RCT will provide evidence for the development of guidelines for the follow-up of LPTB infants in the first 6 months of life to reduce complications, readmissions and developmental problems.

The results of this study can be generalized to tertiary care and community hospitals and the general population.

DETAILED DESCRIPTION:
Late preterm births comprise 70-75% of all preterm births in Ontario and 5.8% of all births in the province. These infants are at significant risk for complications but no guidelines or follow-up programmes exist for decreasing the short and long-term complications associated with LPTB. This project will lay the groundwork for gathering the research evidence to support:

1. An RCT that will study if a specialized LPTB clinic is effective in reducing short-term medical and developmental complications and hospital readmissions,
2. Development of a sustainable long-term follow-up programme supported by evidence,
3. Development of a database to track long-term complications, with the goal of identifying potential risk factors earlier in late preterm infants,
4. Creation and dissemination of Evidence-Based Guidelines, research results for frontline health care providers (GPs, Midwives, etc.), community hospitals and Local Health Integration Networks,
5. Creation and dissemination of Parent Educational Resources for discharge of LPTB infants.

ELIGIBILITY:
Inclusion Criteria:

- singleton or twins born at 34 and 0 days to 36 weeks and 6 days gestational age. Infants admitted to the Level 2 Nursery or newborn nursery at McMaster Children's Hospital or St. Joseph's Healthcare Hamilton or Level 3 Nursery (NICU) at McMaster Children's Hospital will be included.

Exclusion Criteria:

* triplets and infants with major cardiac anomalies, metabolic disorders, significant gastrointestinal anomalies, intrauterine growth restriction, potential genetic syndromes, neurologic anomalies or severe sepsis/meningitis and LPTB requiring mechanical ventilation (post-delivery room resuscitation with prolonged CPAP or intubation) will be excluded.
* mothers who have a history of substance use at any time during pregnancy or alcohol use after confirmation of pregnancy
* participants must be able to understand English and speak English as this pilot does not currently have the financial support to sponsor interpreters.

Max Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 14 months
  Recruitment Rate during first six months of pilot. Reported as the percentage of subjects recruited from those eligible to participate.

SECONDARY OUTCOMES:
Infant Weight Gain | 14 months
  Weight Gain reported in grams.

OTHER OUTCOMES:
Hospital Readmission | 14 months
  The rates of hospital readmission will be determined for the first six months of life.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Giglia, MD FRCP(C) MSc, Principal Investigator — McMaster Children's Hospital & St. Joseph's Hospital
Locations (2):
- Canada (2):
  - St. Joseph's Hospital, Hamilton, Ontario
  - McMaster Children's Hospital & McMaster University, Hamilton, Ontario